CLINICAL TRIAL: NCT02229396
Title: A 28-week, Multicenter, Randomized, Double-Blind, Active-Controlled, Phase 3 Study With a 24-week Extension Phase Followed by a 52-week Extension Phase to Evaluate the Efficacy and Safety of Simultaneous Administration of Exenatide Once Weekly 2 mg and Dapagliflozin Once Daily 10 mg Compared to Exenatide Once Weekly 2 mg Alone and Dapagliflozin Once Daily 10 mg Alone in Patients With Type 2 Diabetes Who Have Inadequate Glycemic Control on Metformin
Brief Title: Phase 3 28-Week Study With 24-Week and 52-week Extension Phases to Evaluate Efficacy and Safety of Exenatide Once Weekly and Dapagliflozin Versus Exenatide and Dapagliflozin Matching Placebo
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: D5553C00003; 2014-003503-29 (EudraCT Number)
Record Dates: First submitted 2014-08-28; First posted 2014-09-01 (Estimated); Results first posted 2017-09-08 (Actual); Last update posted 2018-12-31 (Actual); Status verified 2018-12

CONDITIONS: Diabetes Mellitus
Keywords: Diabetes Mellitus; Exenatide; Dapagliflozin; Diabetes medication; Treatment efficacy; Placebo; Metabolism; Cardiovascular metabolic
MeSH Terms: conditions — Diabetes Mellitus | interventions — dapagliflozin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Exenatide Once Weekly 2 mg and Dapagliflozin Once Daily 10 mg (Experimental)
  Interventions: Drug: Exantide with Dapagliflozin
- Exenatide Once Weekly 2 mg Alone (Experimental)
  Interventions: Drug: Exentide
- Dapagliflozin Once Daily 10 mg Alone (Active Comparator)
  Interventions: Drug: Dapagliflozin

INTERVENTIONS:
Drug: Exantide with Dapagliflozin — 2 mg weekly suspension injection and 10 mg Dapagliflozin
  Arms: Exenatide Once Weekly 2 mg and Dapagliflozin Once Daily 10 mg
Drug: Exentide — 2 mg
  Arms: Exenatide Once Weekly 2 mg Alone
Drug: Dapagliflozin — 10 mg once daily Dapagliflozin
  Arms: Dapagliflozin Once Daily 10 mg Alone

SUMMARY:
Study D5553C0003 is a 28-week, randomized, double-blind, active-controlled, multicenter, Phase 3 efficacy and safety study with 24-week and 52-week extension phases of simultaneous administration of exenatide once weekly (EQW) 2 mg and dapagliflozin 10 mg once daily (QD) compared to EQW 2 mg alone and dapagliflozin 10 mg QD alone in patients with Type 2 diabetes who have inadequate glycemic control on metformin.

ELIGIBILITY:
Inclusion criteria

* Has a diagnosis of T2DM.
* Has HbA1c of 8.0% to 12.0%, inclusive, at Visit 1 and Visit 2.
* Treated with a stable dose of metformin ≥1500 mg/day for at least 2 months prior to Screening.

Exclusion criteria

* FPG ≥280 mg/dL (15.6 mmol/L).
* Serum calcitonin concentration ≥40 pg/mL (≥40 ng/L) at Visit 1 (Screening)
* Clinically significant abnormal free T4 values or patients needing initiation or adjustment of thyroid treatment according to the investigator.
* Abnormal thyroid stimulating hormone (TSH) value at Screening will be further evaluated by free T4.Patients with clinically significant abnormal free T4 values will be excluded.
* Known active proliferative retinopathy.
* History of, or currently have, acute or chronic pancreatitis, or have triglyceride concentrations ≥500 mg/dL (≥5.65 mmol/L) at Visit 1
* History or presence of inflammatory bowel disease or other severe GI diseases, particularly those which may impact gastric emptying, such as gastroparesis or pyloric stenosis.
* History of gastric bypass surgery or gastric banding surgery, or either procedure is planned during the time period of the study. Current use of gastric balloons is also excluded.

Ages: 18 Years to 130 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 695 (Actual)
Dates: Start 2014-09-04 (Actual); Primary Completion 2016-04-26 (Actual); Study Completion 2017-12-28 (Actual)

CONTACTS AND LOCATIONS:
Locations (111):
- United States (64):
  - Research Site, Birmingham, Alabama
  - Research Site, Huntsville, Alabama
  - Research Site, Tuscumbia, Alabama
  - Research Site, Glendale, Arizona
  - Research Site, Tempe, Arizona
  - Research Site, Anaheim, California
  - Research Site, Chula Vista, California
  - Research Site, El Cajon, California
  - Research Site, Fresno, California
  - Research Site, La Mesa, California
  - Research Site, Long Beach, California
  - Research Site, Los Angeles, California
  - Research Site, Mission Hills, California
  - Research Site, Montclair, California
  - Research Site, Oceanside, California
  - Research Site, San Diego, California
  - Research Site, Tustin, California
  - Research Site, Van Nuys, California
  - Research Site, Boynton Beach, Florida
  - Research Site, Clearwater, Florida
  - Research Site, Coral Gables, Florida
  - Research Site, Fort Lauderdale, Florida
  - Research Site, Hialeah, Florida
  - Research Site, Jacksonville, Florida
  - Research Site, Miami, Florida
  - Research Site, North Miami Beach, Florida
  - Research Site, Orlando, Florida
  - Research Site, Tampa, Florida
  - Research Site, Williston, Florida
  - Research Site, Chicago, Illinois
  - Research Site, Avon, Indiana
  - Research Site, Evansville, Indiana
  - Research Site, Franklin, Indiana
  - Research Site, Muncie, Indiana
  - Research Site, Newton, Kansas
  - Research Site, Monroe, Louisiana
  - Research Site, Hazelwood, Missouri
  - Research Site, Bellevue, Nebraska
  - Research Site, Las Vegas, Nevada
  - Research Site, Haddon Heights, New Jersey
  - Research Site, Burlington, North Carolina
  - Research Site, Greensboro, North Carolina
  - Research Site, Mooresville, North Carolina
  - Research Site, Morehead City, North Carolina
  - Research Site, Cincinnati, Ohio
  - Research Site, Vandalia, Ohio
  - Research Site, Medford, Oregon
  - Research Site, Philadelphia, Pennsylvania
  - Research Site, Charleston, South Carolina
  - Research Site, Greer, South Carolina
  - Research Site, Spartanburg, South Carolina
  - Research Site, Summerville, South Carolina
  - Research Site, Dakota Dunes, South Dakota
  - Research Site, Memphis, Tennessee
  - Research Site, Dallas, Texas
  - Research Site, Houston, Texas
  - Research Site, Pearland, Texas
  - Research Site, San Antonio, Texas
  - Research Site, Tomball, Texas
  - Research Site, Clinton, Utah
  - Research Site, Salt Lake City, Utah
  - Research Site, Burke, Virginia
  - Research Site, Manassas, Virginia
  - Research Site, Richmond, Virginia
- Hungary (15):
  - Research Site, Baja
  - Research Site, Balatonfüred
  - Research Site, Budaörs
  - Research Site, Budapest
  - Research Site, Debrecen
  - Research Site, Eger
  - Research Site, Gödöllő
  - Research Site, Gyula
  - Research Site, Kecskemét
  - Research Site, Komárom
  - Research Site, Létavértes
  - Research Site, Nyíregyháza
  - Research Site, Pécs
  - Research Site, Szeged
  - Research Site, Szekszárd
- Poland (7):
  - Research Site, Lodz
  - Research Site, Lublin
  - Research Site, Oświęcim
  - Research Site, Parczew
  - Research Site, Poznan
  - Research Site, Torun
  - Research Site, Zgierz
- Romania (6):
  - Research Site, Baia Mare
  - Research Site, Bucharest
  - Research Site, Galati
  - Research Site, Oradea
  - Research Site, Ploieşti
  - Research Site, Timișoara
- Slovakia (11):
  - Research Site, Banská Bystrica
  - Research Site, Bardejov
  - Research Site, Bratislava
  - Research Site, Dolný Kubín
  - Research Site, Košice
  - Research Site, Levice
  - Research Site, Lučenec
  - Research Site, Nitra
  - Research Site, Pezinok
  - Research Site, Štúrovo
  - Research Site, Trebišov
- South Africa (8):
  - Research Site, Bloemfontein
  - Research Site, Cape Town
  - Research Site, Johannesburg
  - Research Site, Kempton Park
  - Research Site, Middelburg
  - Research Site, Parow
  - Research Site, Port Elizabeth
  - Research Site, Pretoria

REFERENCES:
- [Derived] Jabbour SA, Frias JP, Ahmed A, Hardy E, Choi J, Sjostrom CD, Guja C. Efficacy and Safety Over 2 Years of Exenatide Plus Dapagliflozin in the DURATION-8 Study: A Multicenter, Double-Blind, Phase 3, Randomized Controlled Trial. Diabetes Care. 2020 Oct;43(10):2528-2536. doi: 10.2337/dc19-1350. Epub 2020 Aug 18. PMID 32816874
- [Derived] Guja C, Frias JP, Suchower L, Hardy E, Marr G, Sjostrom CD, Jabbour SA. Safety and Efficacy of Exenatide Once Weekly in Participants with Type 2 Diabetes and Stage 2/3 Chronic Kidney Disease. Diabetes Ther. 2020 Jul;11(7):1467-1480. doi: 10.1007/s13300-020-00815-z. Epub 2020 Apr 18. PMID 32306296
- [Derived] Jabbour SA, Frias JP, Hardy E, Ahmed A, Wang H, Ohman P, Guja C. Safety and Efficacy of Exenatide Once Weekly Plus Dapagliflozin Once Daily Versus Exenatide or Dapagliflozin Alone in Patients With Type 2 Diabetes Inadequately Controlled With Metformin Monotherapy: 52-Week Results of the DURATION-8 Randomized Controlled Trial. Diabetes Care. 2018 Oct;41(10):2136-2146. doi: 10.2337/dc18-0680. Epub 2018 Aug 6. PMID 30082326
- [Derived] Frias JP, Guja C, Hardy E, Ahmed A, Dong F, Ohman P, Jabbour SA. Exenatide once weekly plus dapagliflozin once daily versus exenatide or dapagliflozin alone in patients with type 2 diabetes inadequately controlled with metformin monotherapy (DURATION-8): a 28 week, multicentre, double-blind, phase 3, randomised controlled trial. Lancet Diabetes Endocrinol. 2016 Dec;4(12):1004-1016. doi: 10.1016/S2213-8587(16)30267-4. Epub 2016 Sep 16. PMID 27651331
- See also: CSP_radacted — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_7111&studyid=3057&filename=d5553c00003_revised_csp_3_Redacted.pdf

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study conducted between 04 September 2014 and 28 December 2017. 118 centers in 6 countries randomized patients in the study. A Primary Analysis was performed following completion of the 28-week Treatment Period with a data cut-off date of 26 April 2016. All Primary and Secondary Outcome measures were reported at the time of the Primary Analysis.
Pre-assignment Details: The study had a Screening Visit, a 1-week placebo Lead-in Period, a Randomization Visit, and 9 further visits at 1- to 4-week intervals during a 28-week Treatment Period. Patients then entered a 24-week Extension Period 1 and subsequent 52-week Extension Period 2. A follow-up visit occurred 10 weeks after last dose of study medication.
Groups:
- Dapagliflozin + Placebo: Dapagliflozin 10 milligram (mg) tablet administered orally once daily + matching placebo for exenatide administered as subcutaneous (SC) injection once weekly. Patients continued to administer the same type and dose of metformin therapy they were using at study entry.
- Exenatide + Dapagliflozin: Exenatide once weekly (EQW) 2 mg administered as SC injection + dapagliflozin 10 mg tablet administered orally once daily. Patients continued to administer the same type and dose of metformin therapy they were using at study entry.
- Exenatide + Placebo: Exenatide once weekly (EQW) 2 mg administered as SC injection + matching placebo for dapagliflozin tablet administered orally once daily. Patients continued to administer the same type and dose of metformin therapy they were using at study entry.
Period: Overall Study
Arm/Group | Dapagliflozin + Placebo | Exenatide + Dapagliflozin | Exenatide + Placebo
Started | 233 | 231 | 231
Randomization Code Allocated | 233 | 231 | 231
Safety Analysis Set | 233 | 231 | 230
Intent-to-Treat (ITT) Analysis Set | 230 | 228 | 227
Completed 28-Week Study Period | 208 | 202 | 193
Completed 52-Week Study Period | 194 | 193 | 177
Completed (Completed 104-Week Study Period) | 155 | 154 | 136
Not Completed | 78 | 77 | 95
Not completed — Adverse Event | 6 | 12 | 12
Not completed — Death | 2 | 3 | 1
Not completed — Lost to Follow-up | 14 | 14 | 21
Not completed — Protocol Violation | 2 | 1 | 0
Not completed — Patient Incorrectly Randomized | 0 | 0 | 1
Not completed — Other | 10 | 18 | 15
Not completed — Withdrawal by Subject | 42 | 28 | 41
Not completed — Study-Specific Withdrawal Criteria | 0 | 1 | 3
Not completed — Withdrew; No Record on Termination Page | 2 | 0 | 1

BASELINE CHARACTERISTICS:
Population: The overall number of baseline participants is comprised of the ITT analysis set, defined as all randomized patients who received at least 1 dose of study medication and had at least 1 post-baseline hemoglobin A1c (HbA1c) assessment.
Groups:
- Dapagliflozin + Placebo: Dapagliflozin 10 mg tablet administered orally once daily + matching placebo for exenatide administered as SC injection once weekly. Patients continued to administer the same type and dose of metformin therapy they were using at study entry.
- Total: Total of all reporting groups
Arm/Group | Dapagliflozin + Placebo | Exenatide + Dapagliflozin | Exenatide + Placebo | Total
Number analyzed (Participants) | 230 | 228 | 227 | 685
Age, Continuous [Mean (Standard Deviation); unit: Years] | 54.5 (9.16) [28 to 75] | 53.8 (9.82) [26 to 80] | 54.2 (9.62) [29 to 80] | 54.2 (9.53) [26 to 80]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 120 | 126 | 111 | 357
  Male | 110 | 102 | 116 | 328
Race/Ethnicity, Customized [Number; unit: Participants]
  American Indian Or Alaska Native | 0 | 0 | 2 | 2
  Asian | 1 | 3 | 1 | 5
  Black Or African American | 33 | 34 | 27 | 94
  Other | 7 | 1 | 3 | 11
  White | 189 | 190 | 194 | 573

OUTCOME MEASURES:

1. Primary Outcome: Change in HbA1c From Baseline to Week 28
Description: To compare the change from baseline to Week 28 in HbA1c between exenatide once weekly (EQW) 2 mg and dapagliflozin 10 mg administered simultaneously compared to EQW 2 mg alone and dapagliflozin 10 mg alone.
Time Frame: Baseline to Week 28
Population: The ITT analysis set included all randomized patients who received at least 1 dose of study medication and had at least 1 post-baseline HbA1c assessment.
Measure: Least Squares Mean (95% Confidence Interval); unit: % HbA1c
Arm/Group | Dapagliflozin + Placebo | Exenatide + Dapagliflozin | Exenatide + Placebo
Number analyzed (Participants) | 230 | 228 | 227
% HbA1c | -1.39 [-1.57 to -1.21] | -1.98 [-2.16 to -1.79] | -1.60 [-1.79 to -1.41]
Statistical Analysis 1: Comparison: Exenatide + Dapagliflozin vs Exenatide + Placebo; Test type: Superiority or Other; p = 0.003, Mixed Models Analysis; Treatment, region, baseline HbA1c stratum (<9.0% or ≥9.0%), week, and treatment by week interaction as fixed factors; baseline value as covariate; Mean Difference (Final Values) = -0.38, 95% CI 2-sided [-0.63 to -0.13], Standard Error of Mean 0.129
Statistical Analysis 2: Comparison: Dapagliflozin + Placebo vs Exenatide + Dapagliflozin; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -0.59, 95% CI 2-sided [-0.84 to -0.34], Standard Error of Mean 0.127

2. Secondary Outcome: Change in Body Weight From Baseline to Week 28
Description: To compare the change from baseline to Week 28 in body weight between exenatide once weekly (EQW) 2 mg and dapagliflozin 10 mg administered simultaneously compared to EQW 2 mg alone and dapagliflozin 10 mg alone.
Time Frame: Baseline to Week 28
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: kilogram
Arm/Group | Dapagliflozin + Placebo | Exenatide + Dapagliflozin | Exenatide + Placebo
Number analyzed (Participants) | 230 | 228 | 227
kilogram | -2.22 [-2.78 to -1.66] | -3.55 [-4.12 to -2.99] | -1.56 [-2.13 to -0.98]
Statistical Analysis 1: Comparison: Exenatide + Dapagliflozin vs Exenatide + Placebo; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -2.00, 95% CI 2-sided [-2.79 to -1.20], Standard Error of Mean 0.406
Statistical Analysis 2: Comparison: Dapagliflozin + Placebo vs Exenatide + Dapagliflozin; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -1.33, 95% CI 2-sided [-2.12 to -0.55], Standard Error of Mean 0.400

3. Secondary Outcome: Change in Fasting Plasma Glucose From Baseline to Week 28
Description: To compare the change from baseline to Week 28 in fasting plasma glucose between exenatide once weekly (EQW) 2 mg and dapagliflozin 10 mg administered simultaneously compared to EQW 2 mg alone and dapagliflozin 10 mg alone.
Time Frame: Baseline to Week 28
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: milligrams/deciliter (mg/dL)
Arm/Group | Dapagliflozin + Placebo | Exenatide + Dapagliflozin | Exenatide + Placebo
Number analyzed (Participants) | 230 | 228 | 227
milligrams/deciliter (mg/dL) | -49.19 [-54.91 to -43.47] | -65.83 [-71.60 to -60.06] | -45.75 [-51.67 to -39.83]
Statistical Analysis 1: Comparison: Exenatide + Dapagliflozin vs Exenatide + Placebo; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -20.08, 95% CI 2-sided [-27.95 to -12.20], Standard Error of Mean 4.007
Statistical Analysis 2: Comparison: Dapagliflozin + Placebo vs Exenatide + Dapagliflozin; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -16.64, 95% CI 2-sided [-24.39 to -8.89], Standard Error of Mean 3.947

4. Secondary Outcome: Change From Baseline to Week 28 in 2-hour Postprandial Glucose After a Standard Meal Tolerance Test
Description: To compare the change from baseline to Week 28 in 2-hour postprandial glucose after a standard Meal Tolerance Test between exenatide once weekly (EQW) 2 mg and dapagliflozin 10 mg administered simultaneously compared to EQW 2 mg alone and dapagliflozin 10 mg alone.
Time Frame: Baseline to Week 28
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: mg/dL
Arm/Group | Dapagliflozin + Placebo | Exenatide + Dapagliflozin | Exenatide + Placebo
Number analyzed (Participants) | 230 | 228 | 227
mg/dL | -61.05 [-69.10 to -53.00] | -87.83 [-95.83 to -79.84] | -60.09 [-68.48 to -51.71]
Statistical Analysis 1: Comparison: Exenatide + Dapagliflozin vs Exenatide + Placebo; Test type: Superiority or Other; p < 0.001, ANCOVA; Treatment, region, and baseline HbA1c stratum (<9.0% or ≥9.0%), as fixed factors; baseline value as covariate; Mean Difference (Final Values) = -27.74, 95% CI 2-sided [-37.89 to -17.59], Standard Error of Mean 5.168
Statistical Analysis 2: Comparison: Dapagliflozin + Placebo vs Exenatide + Dapagliflozin; Test type: Superiority or Other; p < 0.001, ANCOVA; Treatment, region, and baseline HbA1c stratum (<9.0% or ≥9.0%), as fixed factors; baseline value as covariate; Mean Difference (Final Values) = -26.78, 95% CI 2-sided [-36.78 to -16.78], Standard Error of Mean 5.090

5. Secondary Outcome: Percentage of Patients Achieving Weight Loss ≥5.0% at Week 28
Description: To compare the percentage of patients achieving weight loss ≥5.0% at 28 weeks between exenatide once weekly (EQW) 2 mg and dapagliflozin 10 mg administered simultaneously compared to EQW 2 mg alone and dapagliflozin 10 mg alone.
Time Frame: Baseline to Week 28
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: % of patients
Arm/Group | Dapagliflozin + Placebo | Exenatide + Dapagliflozin | Exenatide + Placebo
Number analyzed (Participants) | 230 | 228 | 227
% of patients | 20.0 [14.8 to 25.2] | 33.3 [27.2 to 39.5] | 13.7 [9.2 to 18.1]
Statistical Analysis 1: Comparison: Exenatide + Dapagliflozin vs Exenatide + Placebo; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel; Stratified by baseline HbA1c (<9.0% or ≥9.0%); Difference in percentages = 19.7
Statistical Analysis 2: Comparison: Dapagliflozin + Placebo vs Exenatide + Dapagliflozin; Test type: Superiority or Other; p = 0.001, Cochran-Mantel-Haenszel; Stratified by baseline HbA1c (<9.0% or ≥9.0%); Difference in percentages = 13.3

6. Secondary Outcome: Change in Fasting Plasma Glucose From Baseline to Week 2
Description: To compare the change from baseline to Week 2 in fasting plasma glucose between exenatide once weekly (EQW) 2 mg and dapagliflozin 10 mg administered simultaneously compared to EQW 2 mg alone and dapagliflozin 10 mg alone.
Time Frame: Baseline to Week 2
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: mg/dL
Arm/Group | Dapagliflozin + Placebo | Exenatide + Dapagliflozin | Exenatide + Placebo
Number analyzed (Participants) | 230 | 228 | 227
mg/dL | -26.31 [-31.42 to -21.20] | -41.34 [-46.48 to -36.20] | -21.08 [-26.29 to -15.86]
Statistical Analysis 1: Comparison: Exenatide + Dapagliflozin vs Exenatide + Placebo; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -20.26, 95% CI 2-sided [-27.12 to -13.40], Standard Error of Mean 3.494
Statistical Analysis 2: Comparison: Dapagliflozin + Placebo vs Exenatide + Dapagliflozin; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis — This is a nominal p-value; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -15.03, 95% CI 2-sided [-21.85 to -8.20], Standard Error of Mean 3.477

7. Secondary Outcome: Percentage of Patients Achieving HbA1c <7% at Week 28
Description: To compare the percentage of patients achieving HbA1c <7% at 28 weeks between exenatide once weekly (EQW) 2 mg and dapagliflozin 10 mg administered simultaneously compared to EQW 2 mg alone and dapagliflozin 10 mg alone.
Time Frame: Baseline to Week 28
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: % of patients
Arm/Group | Dapagliflozin + Placebo | Exenatide + Dapagliflozin | Exenatide + Placebo
Number analyzed (Participants) | 230 | 228 | 227
% of patients | 19.1 [14.1 to 24.2] | 44.7 [38.3 to 51.2] | 26.9 [21.1 to 32.6]
Statistical Analysis 1: Comparison: Exenatide + Dapagliflozin vs Exenatide + Placebo; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel; Stratified by baseline HbA1c (<9.0% or ≥9.0%); Difference in percentages = 17.9
Statistical Analysis 2: Comparison: Dapagliflozin + Placebo vs Exenatide + Dapagliflozin; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel; Stratified by baseline HbA1c (<9.0% or ≥9.0%); Difference in percentages = 25.6

8. Secondary Outcome: Change in Systolic Blood Pressure From Baseline to Week 28
Description: To compare the change from baseline to Week 28 in systolic blood pressure between exenatide once weekly (EQW) 2 mg and dapagliflozin 10 mg administered simultaneously compared to EQW 2 mg alone and dapagliflozin 10 mg alone.
Time Frame: Baseline to Week 28
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: millimeters of mercury (mmHg)
Arm/Group | Dapagliflozin + Placebo | Exenatide + Dapagliflozin | Exenatide + Placebo
Number analyzed (Participants) | 230 | 228 | 227
millimeters of mercury (mmHg) | -1.8 [-3.4 to -0.3] | -4.3 [-5.8 to -2.7] | -1.2 [-2.8 to 0.4]
Statistical Analysis 1: Comparison: Exenatide + Dapagliflozin vs Exenatide + Placebo; Test type: Superiority or Other; p = 0.005, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -3.0, 95% CI 2-sided [-5.2 to -0.9], Standard Error of Mean 1.08
Statistical Analysis 2: Comparison: Dapagliflozin + Placebo vs Exenatide + Dapagliflozin; Test type: Superiority or Other; p = 0.022, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -2.4, 95% CI 2-sided [-4.5 to -0.4], Standard Error of Mean 1.06

ADVERSE EVENTS:
Time Frame: From baseline (Day 1) up to Week 104 (28-week Treatment Period + 24-week Extension Period 1 + 52-week Extension Period 2).
Description: Treatment-emergent adverse event data is reported for the Safety Analysis set defined as all randomized patients receiving at least 1 dose of study medication. One patient who was randomized did not receive study medication (the patient was randomized in error); this patient was not counted as completing or discontinuing treatment.
Arm/Group | Dapagliflozin + Placebo | Exenatide + Dapagliflozin | Exenatide + Placebo
All-Cause Mortality (participants affected / at risk) | 2/233 | 3/231 | 1/230
Serious Adverse Events (participants affected / at risk) | 18/233 | 17/231 | 18/230
Other Adverse Events (participants affected / at risk) | 73/233 | 87/231 | 78/230
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dapagliflozin + Placebo (N=233) | Exenatide + Dapagliflozin (N=231) | Exenatide + Placebo (N=230)
Abdominal pain lower (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Rib fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Splenic rupture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Acute myocardial infarction (Cardiac disorders) | 2 (2) | 0 (0) | 1 (1)
Angina pectoris (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Arteriosclerosis coronary artery (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 0 (0) | 2 (2)
Bradycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Coronary artery occlusion (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Myocardial infarction (Cardiac disorders) | 0 (0) | 0 (0) | 2 (2)
Palpitations (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Tachycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Tinnitus (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0)
Pituitary-dependent Cushing's syndrome (Endocrine disorders) | 0 (0) | 1 (1) | 0 (0)
Anal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Colitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Gastritis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Pancreatic necrosis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Umbilical hernia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Chest pain (General disorders) | 1 (1) | 0 (0) | 1 (1)
Non-cardiac chest pain (General disorders) | 1 (1) | 0 (0) | 0 (0)
Biliary dyskinesia (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 0 (0) | 2 (2) | 1 (1)
Anaphylactic reaction (Immune system disorders) | 1 (1) | 0 (0) | 1 (1)
Cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (2)
Diverticulitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Meningitis viral (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Osteomyelitis (Infections and infestations) | 1 (2) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Multiple injuries (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Spinal compression fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Toxicity to various agents (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Hepatic enzyme increased (Investigations) | 0 (0) | 0 (0) | 2 (2)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Exostosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Periarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Adenocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Lipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Renal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Diabetic neuropathy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Haemorrhagic stroke (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Ischaemic stroke (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1)
Optic neuritis (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Presyncope (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Transient ischaemic attack (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Suicidal ideation (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Hydronephrosis (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0) | 0 (0)
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dapagliflozin + Placebo (N=233) | Exenatide + Dapagliflozin (N=231) | Exenatide + Placebo (N=230)
Diarrhoea (Gastrointestinal disorders) | 11 (14) | 13 (17) | 17 (25)
Nausea (Gastrointestinal disorders) | 10 (12) | 13 (14) | 26 (29)
Vomiting (Gastrointestinal disorders) | 7 (7) | 8 (10) | 12 (15)
Injection site nodule (General disorders) | 13 (22) | 20 (40) | 14 (24)
Nasopharyngitis (Infections and infestations) | 12 (15) | 15 (17) | 8 (10)
Upper respiratory tract infection (Infections and infestations) | 22 (25) | 15 (22) | 17 (29)
Urinary tract infection (Infections and infestations) | 16 (23) | 19 (31) | 15 (24)
Headache (Nervous system disorders) | 12 (12) | 16 (18) | 12 (12)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
At least 30 days prior to submission for publication or presentation, Authors shall provide Sponsor with such material for its review. Sponsor shall have 30 days to comment. If requested by Sponsor, Authors shall withhold material for an additional 90 days to allow for the taking of measures to establish its proprietary rights. No publication or presentation shall be made unless and until any information determined at Sponsor's sole discretion to be Confidential has been removed.